CLINICAL TRIAL: NCT01019395
Title: An Evaluation of the Pharmacokinetic Profile and Safety of a Single Dose of Daptomycin in Pediatric Subjects Aged 3 Months to Twenty-Four Months Who Are Concurrently Receiving Standard Antibiotic Therapy for Proven or Suspected Bacterial Infection Including Peri-Operative Prophylactic Use of Antibiotics
Brief Title: Pharmacokinetics (PK) and Safety Evaluation of Daptomycin in Children Ages 3-24 Months With Proven or Suspected Gram-positive Infections or Peri-Operative Subjects Receiving Prophylactic Antibiotics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3009-018; DAP-PEDS-09-01 (Other: Cubist Study Number)
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Gram Positive Bacterial Infection
Keywords: Gram Positive Infection; Concurrent Antibiotic Treatment
MeSH Terms: conditions — Gram-Positive Bacterial Infections | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Group 1: Ages 13 months to 24 months inclusive. Six subjects dosed at 6 mg/kg as a 30 minute infusion.
  Interventions: Drug: Daptomycin
- Group 2 (Experimental): Group 2: Ages 7 months to 12 months inclusive: Six subjects will receive a dose of 4 mg/kg as a 30 minute infusion
  Interventions: Drug: Daptomycin
- Group 3 (Experimental): Group 3: Ages 3 months to 6 months inclusive: Six subjects will receive a dose of 4 mg/kg as a 30 minute infusion.
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — Group 1: Ages 13 months to 24 months inclusive. Six subjects dosed at 6 mg/kg as a 30 minute infusion;
  Group 2:Ages 7 months to 12 months inclusive: Six subjects will receive a dose of 4 mg/kg as a 30 minute infusion;
  Group 3: Ages 3 months to 6 months inclusive: Six subjects will receive a dose of 4 mg/kg as a 30 minute infusion.
  Other Names: Cubicin

SUMMARY:
This is a research study designed to look at the pharmacokinetics (distribution, breakdown, and removal) and tolerability of a single dose of daptomycin in patients aged 3 months to 24 months who have proven or suspected infections that are caused by a specific group of bacteria (called Gram-positive bacteria)or perioperative subjects that are receiving prophylactic antibiotics .

ELIGIBILITY:
Inclusion Criteria:

1. Written parental (or appropriate legal representative) informed consent prior to any study-related procedure not part of normal medical care; 2.1 Male or female between the ages of 3 months and 24 months, inclusive; 3. Able to comply with the protocol for the duration of the study; 4.1 Clinically stable with no evidence of hemodynamic instability (defined as a requirement for inotropic or vasodilatory support to manage blood pressure) in the 24 hour window prior to first dose, and no history or evidence of renal or hepatic compromise; 5.1 Suspected or diagnosed bacterial infection for which the subject is receiving standard antibiotic therapy; including prophylactic use of antibiotics peri-operatively; 6. A calculated creatinine clearance rate (CLcr) ≥ 80 ml/min/1.73m2 as determined by the Schwartz equation at baseline; 7. Creatine phosphokinase (CPK) levels less than 2X ULN (upper limit of normal) at baseline; 8.1 Presence of two patent intravenous lines (or comparable means of venous or arterial access)prior to dosing on Study Day 1. A single intravenous line (or comparable means of venous access) is acceptable for both drug administration and sample collection if reasonable effort to gain a second line is unsuccessful. The line must be flushed as described in Appendix B of the protocol prior to obtaining PK samples. PK sample can be obtained from a peri-operatively placed arterial line. Arterial PK samples should be indicated on the CRF.

Exclusion Criteria:

1. Investigational drug use (including daptomycin) or participation in any experimental procedure in the 30 days preceding study entry;
2. Known allergy/ hypersensitivity to daptomycin; 3.1 History of clinically significant, renal, hepatic, autoimmune disease or primary immune deficiency;

4. Deleted 5. Subjects with clinically significant abnormal laboratory test results (including ECGs), as determined by Investigator; 6. Administration of rifampin within 7 days of study drug administration; 7. Deleted 8. Subjects in whom collection of the required blood volume would put them at risk of hemodynamic disturbance (at the discretion of Investigator); 9. Deleted; 10.1 Planned administration of intramuscular injection within 12 hours following study administration unless approved by the Medical Monitor; 11. Deleted 12.1 Guillian-Barre or spinal cord injury; 13. History of or current rhabdomyolysis.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2010-01-05 (Actual); Primary Completion 2012-03-20 (Actual); Study Completion 2012-03-20 (Actual)

PRIMARY OUTCOMES:
PK of single dose daptomycin in subjects between 3 and 24 months who are receiving standard antibiotic therapy for a Gram-positive infection, including subjects that are receiving prophylactic antibiotics peri-operatively. | Two years

SECONDARY OUTCOMES:
Safety of a single dose daptomycin in subjects between 3 and 24 months, who are receiving standard antibiotic therapy for a Gram-positive infection, including subjects that are receiving prophylactic antibiotics peri-operatively. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Paula Bokesch, MD, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (8):
- United States (8):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital-San Diego, San Diego, California
  - University of Louisiana at Monroe, Shreveport, Louisiana
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - Cook Children's Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Bradley JS, Benziger D, Bokesch P, Jacobs R. Single-dose pharmacokinetics of daptomycin in pediatric patients 3-24 months of age. Pediatr Infect Dis J. 2014 Sep;33(9):936-9. doi: 10.1097/INF.0000000000000318. PMID 25361023